CLINICAL TRIAL: NCT05855434
Title: Assessing Cognitive Deterioration in COVID-19 (ACDC) Cognitive Impairment After COVID-19 - Inflammatory and Neural Correlates: A Pilot Study
Brief Title: The ACDC Study Assessing Cognitive Deterioration in COVID-19
Acronym: ACDC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Grampian (Other Government)
Collaborators: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS Project ID 314094
Record Dates: First submitted 2023-04-04; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: SARS-CoV-2 Infection; Cognitive Change; Cognitive Dysfunction
MeSH Terms: conditions — COVID-19; Cognitive Dysfunction | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Magnetic Resonance Imaging/Magnetic Resonance Spectroscopy

SUMMARY:
The long-term impact and effects of COVID-19 are still being determined. However, what is clear, is that some people are still struggling following a period of illness with COVID-19. Now known as 'long covid' or 'post covid-19 syndrome', people are not only experiencing physical symptoms like fatigue and breathlessness, but also psychological difficulties, as well as cognitive changes often referred to as 'brain fog'. This can include symptoms, such as changes in memory, difficulties with organisation and problem solving, as well as the ability to concentrate.

Evidence from other research areas suggest that these changes could be due to shrinkage in areas of the brain that control functions like memory and concentration. There are also connections between different brain areas that work together to perform tasks such as remembering and concentrating, and these areas may also be affected by COVID-19.

The purpose of this study is to scan the brains of patients reporting cognitive changes having been hospitalised with COVID-19 infection to see if any of these areas or connections have changed after infection and whether this might explain these cognitive changes.

DETAILED DESCRIPTION:
BACKGROUND OF PROPOSED INVESTIGATION

Overview

A heterogenous cohort of patients, who have been variably denoted as suffering from "Long COVID" or the Post COVID-19 Syndrome, will have persistent cognitive and affective symptoms. A recent large systematic review found that fatigue and objective cognitive impairment were common and persistent after COVID-19 disease with a prevalence of 24.4% and 20.2% respectively (Badenoch et al., 2022). The severity of physical illness associated with SARS-CoV2 infection does not correlate with the likelihood of these symptoms developing or persisting, raising the questions as to the nature of the processes driving post COVID-19 cognitive symptoms.

The effects of COVID-19 disease on the brain and the link to cognitive impairment has been emphasised as an area of priority research (Samkaria and Mandal, 2021). There have been proposed mechanistic explanations from case studies (Yesilkaya et al., 2021) as well as more general commentaries on the neuroimmune correlates of COVID-19 disease, (Yesilkaya and Balcioglu, 2020) but as yet no high-quality evidence exists.

It is suggested that COVID-19 disease may lead to pathologically identifiable brain changes. A large study evaluating structural brain imaging of patients before and after SARS-CoV2 infection using United Kingdom (UK) Biobank data found evidence of grey matter volume reduction compared with controls (Douaud et al., 2022). This mainly involved olfactory areas but wider limbic involvement was discussed in the context of memory impairment and reported cognitive change. A much smaller study (Hosp et al., 2021) correlated functional imaging changes, Fluoro-Deoxy-Glucose Positron Emission Tomography (FDG-PET), with cognitive impairment in patients hospitalised with COVID-19 disease.

Magnetic Resonance Spectroscopy (MRS) is an imaging technology that represents a non-invasive diagnostic tool for evaluating white matter injury in the brain and can provide valuable information regarding underlying pathogenesis. Most importantly, MRS can identify neurochemical abnormalities even in the absence of corresponding findings on structural MR brain imaging. This is important, in that many patients with persistent cognitive symptoms have normal conventional imaging (Hellgren et al., 2021).

MRS has been used in a small preliminary study to outline brain inflammation and damage linked to COVID-19 disease (Rapalino et al., 2021). This work pointed to characteristic white matter inflammatory MRS findings in patients with severe and acute COVID-19 disease. White matter changes have also been described using conventional MR imaging in patients presenting with cognitive impairment in association with COVID-19 disease (Hellgren et al., 2021) but such results were not replicated in patients describing "brain fog" symptoms after hospitalisation for COVID-19 disease (Sklinda et al., 2021).

Reviewing the nascent investigation already undertaken, there is a possibility that inflammation and other neural correlates play a role in persistent cognitive symptoms in those who have been infected with SARS-CoV2. This pilot study aims to investigate these links as a necessary and urgent first step in trying to understand how and why a significant number of patients are affected in this way.

Local relevance

NHS Grampian, along with the other health boards in Scotland, has received funding from the Scottish Government to identify and provide intervention for the mental health needs of patients hospitalised with COVID-19 disease. This follows on from Coronavirus (Covid-19): Mental health needs of hospitalised patients - report (https://www.gov.scot/publications/mental-health-needs-patients-hospitalised-due-covid-19/).

This has been identified as an unmet need and a clinical priority. The response has seen the creation of the Mental Health After Covid-19 Hospitalisation Team (MACH). NHS Grampian is amongst a small leading group of other boards in rolling out this service and clinicians are currently contacting eligible patients to offer screening appointments as well as developing mental health interventions.

NHS Grampian is also moving forward with resources to help staff affected by COVID-19 disease. NHS Grampian's "We Care" programme is expanding to address the identified needs of staff affected by the pandemic, which will include the better identification, understanding and management of 'Long COVID'. There is therefore a significant overlap in the NHS Grampian corporate response for staff and the wider clinical strategy. This underlines the importance and centrality of addressing the longer-term effects of COVID-19 disease for both staff and patients alike.

Embedding research within the scope of the work of the MACH team is very important. There is a lot that remains unknown about the COVID-19 disease and meaningful inquiry about associated long term effects is an important and pressing issue.

Patients suffering with the long-term sequelae of COVID-19 disease will have a range of needs. In particular, a pressing concern for them is cognitive change. Within NHS Grampian there have been reports anecdotally from significant numbers of patients who have been seen in the MACH clinics so far. The prevalence of cognitive change, specifically impaired recall, has been estimated at 25% of patients from 12 to 18 months after SARS-CoV2 infection (Becker et al., 2021). In a recent large meta-analysis it was found that 32% of patients reported fatigue and 22% had evidence of cognitive impairment 12 weeks or more after SARS-CoV2 infection (Ceban et al., 2022).

Investigators plan to offer neuropsychometric testing to all patients who report persistent cognitive symptoms in order to better understand the particular pattern, or phenotype, encountered by patients. It will be important to consider why it is that some patients report prolonged symptoms in general and prolonged cognitive symptoms specifically. Neuroimaging, and spectroscopy specifically, could start to provide answers to these questions.

The proposed project will enable research into a common adverse outcome of COVID-19 disease, which has both national recognition and significant morbidity (Ceban et al., 2022).

ELIGIBILITY:
PARTICIPANTS:

Inclusion Criteria

* A patient who has been hospitalised with COVID-19 disease (with a positive Polymerase Chain Reaction (PCR) result for SARS-CoV2 infection) within NHS Grampian hospitals with subsequent subjective reporting and objective evidence of cognitive change.
* Patients aged over 18.
* Patient has completed neuropsychometric testing protocol as described above.
* Participant who is willing and able to give informed consent for participation in the study.

Exclusion Criteria

* Any patient whose physical condition will preclude them from lying still for the duration of the brain scan.
* Contraindication to magnetic resonance scanning such as an implantable cardiac device.
* Patients who required intensive care treatment for SARS-CoV2 infection.
* Patients with a pre-existing diagnosis of a Neurodegenerative disease (eg. Dementia), Intellectual Disability, previous moderate/severe brain injury or previous brain injury with noted cognitive change.
* Patients with a pre-existing neuro-inflammatory disorder (eg. Multiple Sclerosis).
* Patients under investigation for, or with a history of, cognitive change prior to hospitalisation with COVID-19 disease.
* Patients with a dependency on alcohol or recreational drugs.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 16 and over who were hospitalised due to SARS-CoV-2 infection, having a positive PCR, and reporting cognitive change from baseline in the NHS Grampian region of Scotland.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint The primary endpoint is MR imaging and spectroscopy associations with measured cognitive performance. | June 2024
  To report the association (present or not) between MR imaging and spectroscopy measures and cognitive performance following hospitalisation for COVID-19 disease.

SECONDARY OUTCOMES:
Metabolic profile of selected brain regions via MRS | June 2024
  Magnetic Resonance Spectroscopy reports metabolic profiles of various biochemical processes in the brain.
White matter assessment via Tract Based Spatial Statistics (TBSS) | June 2024
  This is the analysis of diffusion data as it pertains to Brain white matter.
Brain iron levels | June 2024
  Brain Iron levels are a proxy for inflammation and will be assessed in regions reported to be related to memory performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, Grampian, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT05855434/Prot_000.pdf